## **OFFICIAL TITLE OF THE STUDY:**

# EFFECT OF DILUTED THYME HONEY ON DRY MOUTH IN INTENSIVE CARE UNIT PATIENTS EXPOSED TO OXYGEN FLOW THERAPY: A RANDOMIZED CONTROLLED STUDY

**DOCUMENT TYPE: DATA ANALYSIS** 

## **RESEARCHERS:**

- ESRA YAPRAK GÖKTÜRK (MSC)
   ANKARA UNİVERSİTY
  GRADUATE SCHOOL OF HEALT SCİENCES
  - AYTEN DEMİR (PROFESSOR DOCTOR)
    ANKARA UNİVERSİTY
    FACULTY OF NURSING

**DOCUMENT DATE: 30/11/2022** 

**ANKARA/TURKEY** 

## EFFECT OF DILUTED THYME HONEY ON DRY MOUTH IN INTENSIVE CARE UNIT PATIENTS EXPOSED TO OXYGEN FLOW THERAPY: A RANDOMIZED CONTROLLED STUDY

• NCT ID: Not Yet Assigned

### • Correspondance

Esra Yaprak Göktürk (eyk1994.ek@gmail.com) (+905377819714)

## • Esra Yaprak GÖKTÜRK

Nursing Department Thesis Master's Program, Institute of Health Sciences, Ankara University

eyk1994.ek@gmail.com

Clinical Trials Organization: AnkaraU

**Clinical Trials User: EYGokturk** 

### Ayten DEMİR

Faculty of Nursing, Department of Nursing, Ankara University, Ankara Türkiye aytendemirankara@gmail.com

https://orcid.org/0000-0002-5677-2347

#### • Ethics Statement

To conduct this research, ethics committee approval (number 56786525-050.04.04/737202) dated November 30, 2022, was obtained from the Ankara University Rectorate Ethics Committee. Institutional approval (meeting number 0137) dated September 18, 2022, was obtained from the Ankara Training and Research Hospital, where the research was conducted. This study was completed as a master's thesis in the Nursing Department program at Ankara University, Institute of Health Sciences.

## • Data Availability Statement

We have confirmed that the methods used in data analysis are appropriate. They were applied to our data within the study design and context, and the statistical results were applied and interpreted correctly. As a condition of journal submission, we accept responsibility for ensuring that the selection of statistical methods is appropriate and is performed and interpreted correctly. The data and original materials contained in this study can be obtained by contacting Esra Yaprak Göktürk, one of the authors of this study, at eyk1994.ek@gmail.com

#### **DATA ANALYSIS**

The data collected in the study were analyzed using SPSS (Statistical Package for Social Sciences) for Windows 22.0 program. Descriptive statistical methods such as number, percentage, mean, and standard deviation were used to evaluate the data. Differences between the rates of categorical variables in the independent intervention and control groups were analyzed using Chi-Square and Fisher exact tests. Kurtosis and Skewness values were analyzed to determine whether the variables of the study were normally distributed.

Table 1. Normal Distribution of Intensive Care Unit Patients Receiving Nasal Oxygen Flow Therapy in Control and Intervention Groups

| VARIABLES | Control Group (n=32) | | Intervention Group (n=32) | |
|---|---|---|---|---|
| | Kurtosis | Skewness | Kurtosis | Skewness |
| Dry mouth pretest | -1,115 | -0,169 | -0,949 | -0,287 |
| Swallowing difficulty pretest | -1,336 | 0,148 | -1,051 | 0,214 |
| Speech difficulty pretest | -1,445 | 0,165 | -1,222 | 0,273 |
| Pre-test waking up from sleep with dry mouth body | -0,994 | 0,356 | -0,695 | 0,557 |
| Dry tongue pretest | -1,171 | 0,281 | -0,758 | 0,570 |
| Burning in the mouth pretest | -1,261 | -0,009 | -1,223 | 0,018 |
| Preliminary test for dryness in the throat | -0,448 | -0,268 | 1,214 | -1,136 |
| Thirst pre-test | -1,342 | -0,450 | -0,350 | -0,871 |
| Bad taste in the mouth pretest | 0,555 | 0,739 | -0,213 | -0,370 |
| Saliva quantity pretest | -0,339 | -0,412 | -0,319 | -0,677 |
| Pre-test for bad breath odor | -0,032 | 0,525 | -0,398 | 0,501 |
| Dry mouth post-test | -0,464 | -0,660 | -0,906 | -0,084 |
| Swallowing difficulty post-test | -1,544 | 0,141 | -0,724 | -0,062 |
| Speech difficulty post-test | -1,462 | 0,228 | -0,940 | 0,555 |
| Waking up from sleep with dry mouth body post-test | -0,043 | 0,830 | -0,582 | 0,804 |
| Dry tongue post-test | -1,158 | 0,381 | -1,242 | 0,426 |
| Burning in the mouth final test | -0,220 | 0,719 | -1,061 | 0,301 |
| Final test for dryness in the throat | -0,369 | -0,358 | -0,132 | -0,307 |
| Thirst final test | -0,496 | -0,169 | -0,940 | -0,379 |
| The last test of bad taste in the mouth | -0,194 | 0,893 | -0,558 | 0,404 |
| Saliva quantity post-test | -0,352 | 0,241 | 1,154 | -1,321 |
| The last test of bad breath odor | 0,721 | 0,888 | 0,987 | 1,039 |